CLINICAL TRIAL: NCT02559999
Title: Objective Markers of Pain Perception in Humans: a Study in Healthy Subjects
Brief Title: Objective Markers of Pain Perception in Humans
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Saint Etienne (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 1308172; 2013-A01636-39 (Other: ANSM)
Record Dates: First submitted 2015-09-24; First posted 2015-09-25 (Estimated); Last update posted 2018-10-23 (Actual); Status verified 2018-10

CONDITIONS: Healthy
Keywords: Healthy Volunteers; Pain; EEG
MeSH Terms: conditions — Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- EEG responses (Other): The study compares electroencephalographical responses (EEG) to painful stimuli tonic to those evoked by non-painful stimuli and with or without virtual reality
  Interventions: Other: Painful tonic stimuli; Other: non-painful stimuli

INTERVENTIONS:
Other: Painful tonic stimuli
Other: non-painful stimuli

SUMMARY:
Determine objective markers of pain perception remains a major scientific and medical issue. Various tools have been proposed to objectify pain, but their adaptability to different clinical contexts are limited. Our working hypothesis considers that the research for markers of immediate pain perception should be based on an electrophysiological approach, based on the combined analysis of EEG and autonomic responses.

DETAILED DESCRIPTION:
This project aims to study the cortical and autonomic responses induced by tonic painful stimulation compared to those induced by comparable sensory and stressful stimulations, by combining high density EEG, cutaneous sympathetic, cardiovascular and pupillary recordings.

ELIGIBILITY:
Inclusion Criteria:

* Affiliate or beneficiary of social security
* Signature of consent

Exclusion Criteria:

* History of cardiovascular disease (vagal syncope, hypertension, etc ...), renal, metabolic (diabetes ...), psychiatric (depression, etc ...) or neurological (seizure, etc ...) syndromes;
* Reynaud's syndrome;
* Raynaud's disease;
* Acrocyanosis;
* Known rhythm disorders;
* Participation at the same time in another clinical trial;
* Taking a medical treatment;
* Suffering from acute (complaint of pain in the week before the test) or chronic pain,
* Allergic to conductive gel for electrodes.

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 21 (Actual)
Dates: Start 2014-06-04 (Actual); Primary Completion 2018-02-28 (Actual); Study Completion 2018-02-28 (Actual)

PRIMARY OUTCOMES:
EEG Gamma power. | Baseline
  The EGG signals are compared between a painful stimuli tonic to those evoked by non-painful stimuli.

SECONDARY OUTCOMES:
ratio of low to high frequency spectral powers | Baseline
  The low and high frequency spectral powers are measured by an ECG Holter. The ratio are compared between a painful stimuli tonic to those evoked by non-painful stimuli.
Magnitude of the sympathetic cutaneous reactivity | Baseline
  The sympathetic cutaneous reactivity is measured by an acquisition system (ME6000, MEDIMEX, France) with one electrode on the hand.
  The magnitudes are compared between a painful stimuli tonic to those evoked by non-painful stimuli.
Amplitude of pupillary dilation | Baseline
  The pupillary dilation is measured by the ISCAN® system (MA, USA). The amplitudes are compared between a painful stimuli tonic to those evoked by non-painful stimuli.

CONTACTS AND LOCATIONS:
Overall Officials: Roland PEYRON, MD, Principal Investigator — CHU de SAINT-ETIENNE
Locations (2):
- France (2):
  - Hospices Civils de LYON, Lyon
  - CHU de SAINT-ETIENNE, Saint-Etienne

IPD SHARING:
Plan to Share IPD: No